CLINICAL TRIAL: NCT00831701
Title: Medical Expulsive Therapy of Single Distal Ureteral Stones. A Randomised, Double-blind and Placebo-controlled Study
Brief Title: Medical Expulsive Therapy of Single Distal Ureteral Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Räto T. Strebel, Department of Urology, University Hospital Zürich, switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-Hermanns
Record Dates: First submitted 2008-11-19; First posted 2009-01-29 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Ureteral Calculi
Keywords: Adrenergic alpha antagonists; drug therapy; tamsulosin; ureter
MeSH Terms: conditions — Ureteral Calculi | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin (Active Comparator): Tamsulosin treatment
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — 0.4 mg Tamsulosin once daily for 21 days
  Other Names: Pradif; Flomax
  Arms: Tamsulosin
Drug: Placebo — One placebo pill per day for 21 days or until stone expulsion
  Arms: Placebo

SUMMARY:
Current therapeutic options for ureteral stones include active intervention as well as conservative "watch and wait" approaches. Endoscopic treatment of ureteral stones has a high success rate and reliably results in immediate stone removal However, surgical as well as anaesthetic risks are not negligible and serious complications are possible. For many patients, a conservative treatment is an appealing option. Watchful waiting, however, not always results in stone clearance and may be associated with recurrent renal colics.

The therapeutic potential of alpha-blockers for ureteral stone disease has been investigated prompted by the detection of alpha-receptors in ureteral smooth muscle cells. Blocking of such receptors, which are predominantly located in the distal part of the ureter results in relaxation of the ureteral wall and modulation of peristaltic activity. This mechanism has been proposed to facilitate stone passage for ureteral calculi.

Numerous clinical trials have revealed a significant improvement of the stone expulsion rate using the alpha-blocker tamsulosin. Most of these studies were randomised but none were performed in a double-blind and placebo-controlled fashion. Therefore, the objective of this trial was to evaluate the efficacy of medical expulsive therapy with tamsulosin in a randomised, double-blind, placebo-controlled setting.

ELIGIBILITY:
Inclusion criteria:

* patients with a single 2 to 7mm ureteral stone below the common iliac vessels

Exclusion criteria:

* presence of multiple ureteral stones
* renal insufficiency (glomerular filtration rate below 60 ml/min)
* urinary tract infection
* a solitary kidney
* pregnancy
* history of ureteral surgery or previous endoscopic procedure
* hypersensitivity to tamsulosin
* current alpha-blocker, calcium-antagonist or corticosteroid medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Department of Urology, University Hospital Zürich, Switzerland, Zurich, Switzerland

REFERENCES:
- [Derived] Hermanns T, Sauermann P, Rufibach K, Frauenfelder T, Sulser T, Strebel RT. Is there a role for tamsulosin in the treatment of distal ureteral stones of 7 mm or less? Results of a randomised, double-blind, placebo-controlled trial. Eur Urol. 2009 Sep;56(3):407-12. doi: 10.1016/j.eururo.2009.03.076. Epub 2009 Apr 3. PMID 19375849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomisation of 100 pts between 09.2006 and 09.2008 in a University Hospital
Pre-assignment Details: 10 patients were excluded from the final analysis due to stone expulsion before medication intake or withdrew of consent
Groups:
- Tamsulosin Treatment: Patients received one pill of Tamsulosin 400 micrograms once daily
- Placebo Treatment: Patients received Placebo pill once daily
Period: Overall Study
Arm/Group | Tamsulosin Treatment | Placebo Treatment
Started | 50 | 50
Completed | 45 | 45
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Stone expulsion before first medication | 2 | 2
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 45 | 93
  >=65 years | 2 | 5 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.7) | 43.4 (13.9) | 40.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 42 | 39 | 81
Region of Enrollment [Number; unit: participants]
  Switzerland | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stone Expulsion
Description: The primary end point was the number of patients per group experiencing stone expulsion until day 21, as confirmed by low-dose abdominal computed tomography (CT).
Time Frame: 21 days
Measure: Number; unit: Participants
Arm/Group | Tamsulosin Treatment | Placebo Treatment
Number analyzed (Participants) | 45 | 45
Participants | 39 | 40

2. Secondary Outcome: Time to Stone Passage
Description: The patient-defined time of stone expulsion was considered the event for time to stone passage. Patients with unnoticed stone expulsion were censored at the date of last positive stone status, and those who discontinued the therapy were censored at the date of last medication intake. Kaplan-Meier estimates were computed for time to stone passage.
Time Frame: 21 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tamsulosin Treatment | Placebo Treatment
Number analyzed (Participants) | 45 | 45
days | 7 [3 to 10] | 10 [3 to 20]

3. Secondary Outcome: Required Analgesics
Description: Oral diclophenac (up to 3x50 mg pills) as first-line and oral metamizole (up to 8x 500mg pills)as second-line on-demand analgesics were prescribed. All patients were requested to record the required amount of pills per day
Time Frame: Until stone expulsion or up to 21 days
Measure: Median (Inter-Quartile Range); unit: pills per day
Arm/Group | Tamsulosin Treatment | Placebo Treatment
Number analyzed (Participants) | 45 | 45
pills per day | 3 [1 to 9.8] | 7 [4 to 16]

4. Secondary Outcome: Maximum Daily Pain Score
Description: All patients kept a diary to record the score of every painful episode on a 10-cm visual analogue scale (0= no pain at all; 10= strongest pain one can imagine).
Time Frame: Until stone expulsion or up to 21 days
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tamsulosin Treatment | Placebo Treatment
Number analyzed (Participants) | 45 | 45
Units on a scale | 3 [0 to 10] | 7 [0 to 9]

5. Secondary Outcome: Number of Participants Requiring Active Treatment
Description: The number of participants requiring active treatment was recorded. Shock wave lithotrypsy (SWL), ureterorenoscopy (URS) or insertion of an ureteral catheter were considered as active treatment.
Time Frame: 21 days
Measure: Number; unit: participants
Arm/Group | Tamsulosin Treatment | Placebo Treatment
Number analyzed (Participants) | 45 | 45
participants | 6 | 4

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Tamsulosin Treatment | Placebo Treatment
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 4/45 | 1/45
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin Treatment (N=45) | Placebo Treatment (N=45)
Retrograde ejaculation (Reproductive system and breast disorders) | 2 (2) | 0 (0) — R.E. during medication
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cutaneous reaction (mild) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Not all patients were able to record the exact time of stone passage. Thus, the secondary end point of time to stone passage is based on Kaplan-Meier estimation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No